CLINICAL TRIAL: NCT06878274
Title: Radiotherapy to Optimize Event-free Survival Following Chemo-Immunotherapy and Surgery in Upper Stage III NSCLC With Evidence of Pathological Residual Disease (RESCUE): Phase II Trial
Brief Title: Post-operative Radiotherapy After Neodjuvant Chemo-immunotherapy and Surgery in Stage III NSCLC
Acronym: RESCUE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Houda Bahig, Radiation Oncologist, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESCUE
Record Dates: First submitted 2024-12-04; First posted 2025-03-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Non Small Cell Lung Cancer; Stage III Lung Cancer
Keywords: Post operative radiotherapy; lung cancer; non small cell lung cancer; stage III lung cancer; neoadjuvant immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-operative radiotherapy (Experimental): Mediastinal PORT (40 Gy in 15 fractions) within 24 weeks from thoracic surgery
  Interventions: Radiation: Post-operative radiotherapy
- No post-operative radiotherapy (No Intervention): No post-operative radiotherapy (PORT)

INTERVENTIONS:
Radiation: Post-operative radiotherapy — Mediastinal post-operative radiotherapy to a dose of 40 Gy in 15 fractions
  Arms: Post-operative radiotherapy

SUMMARY:
This study investigates whether postoperative radiotherapy (PORT) improves outcomes for patients with stage III non-small cell lung cancer (NSCLC) who have residual disease after neoadjuvant chemo-immunotherapy and surgery. The primary objective is to compare event-free survival (EFS) between patients receiving PORT targeting involved lymph node regions and those without PORT. Secondary and tertiary endpoints include overall survival, locoregional and distant control, toxicity, and quality of life. The phase II randomized trial will enroll 118 patients, stratifying by adjuvant immunotherapy use, with follow-up extending up to 5 years. Statistical analysis aims to detect a 15% improvement in 2-year EFS, with a total study duration of 7 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥ 18 years old
2. Ability to provide written informed consent
3. ECOG performance status 0-2
4. Histologically confirmed NSCLC
5. Absence of actionable driver mutation (EGFR/ALK/ROS)
6. Complete preoperative imaging staging, including: FDG-PET and brain imaging to exclude distant metastases will be mandatory.
7. Baseline clinical or post-operative pathological stage III including specifically stage T1-4N2-3
8. Completion of 2-4 cycles of neoadjuvant chemo-IO, regardless of the specific immunotherapy and chemotherapy used.
9. Status post-complete (R0) surgical resection with mediastinal lymph node dissection.
10. Residual nodal disease on final pathology specimen (i.e. absence of pathological complete response).
11. Postoperative lung function examination: FEV1 > 1 L (or greater than 35% expected value)

Exclusion Criteria:

1. Pregnant individuals
2. Previous chest radiotherapy
3. >24 weeks after thoracic surgery
4. History of other non-cutaneous neoplasms within the last 24 months
5. Active grade ≥ 2 pneumonitis.
6. Presence of interstitial lung disease
7. Recurrence or metastasis occurred
8. Medical conditions that hinders the safe administration of radiotherapy or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | Defined as the time from random assignment to loco-regional or distant recurrence, or death from any cause, assessed up to 60 months.

SECONDARY OUTCOMES:
Overall Survival | Time from random assignment to death from any cause, assessed up to 60 months.
Grade 3 Toxicity | Classified as early (within the first 3 months) or late (after 3 months), assessed up to 60 months.
Locoregional control | Time from random assignment to locoregional recurrence, proven radiologically and/or pathologically, assessed up to 60 months.
Distant metastasis free survival | Time from random assignment to distant recurrence, proven radiologically and/or pathologically, or death from any cause, assessed up to 60 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD includes anonymized individual participant data collected throughout the course of the study and may include the analyzable data set.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: study completion date, up to 60 months.